CLINICAL TRIAL: NCT04348123
Title: A Proposed Community-Based Interventional Program That Educates, Identifies And Overcomes Barriers to Complete Screening Mammography Among Homeless Women
Brief Title: Interventional Program Educates, Identifies + Overcomes Barriers to Complete Screening Mammography
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CASE10119
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Outreach educational program (Experimental): Participants will be given a survey to elucidate beliefs and barriers around breast health and mammography.
  A brief, culturally-appropriate educational session about breast health and mammography will follow and will be delivered by a female public health educator.
  After education, eligible women will be offered a free on-site mammogram
  Interventions: Other: Survey; Behavioral: Education Session

INTERVENTIONS:
Other: Survey — Survey questionnaire seeks to collect data relevant to mammogram completion, barriers, and facilitators
Behavioral: Education Session — After the survey, clinic staff will conduct brief, culturally-appropriate educational session about breast health and mammography delivered by a female public health educator with experience in the underserved community. Educational session will explain screening options and address common barriers

SUMMARY:
The purpose of this study is to identify interventions that are designed to better serve women who are homeless, with a speciﬁc focus on increasing screening rates and decreasing late stage breast cancer diagnosis among this high-risk understudied community of women. As a result, the study team hopes to influence the broader homeless healthcare initiative

DETAILED DESCRIPTION:
The goal of this program will be to bring 6-8 mobile on site mammography clinics to homeless shelters that house women over a two-year period. Prior to arrival, clinic staff will recruit women to participate in a survey to elucidate beliefs and barriers around breast health and mammography. After the survey, clinic staff will conduct the outreach program, consisting of a brief educational session about breast health and mammography for any participating women. Education will be tailored to be culturally appropriate, and delivered by a female public health educator with experience in the underserved community. The educational session will explain screening options and address common barriers. After education, eligible women who wish to receive a mammogram may receive one from the on-site mobile mammography clinic free of charge. Throughout the day, the community educator will also lead activities and meals will be provided in order to create a festive atmosphere and inspire a sense of community among the women. Spanish speaking staff will be available for the educational sessions.

ELIGIBILITY:
Inclusion Criteria:

* Women under age 40 who present with high risk breast cancer related symptoms or a first degree relative with breast cancer
* Have not had mammogram in the last 12 months
* Resident at a homeless shelter or transitioning housing facility.

Exclusion Criteria:

- Participant experiencing homelessness under age 40 who DO NOT present with high risk breast cancer related symptoms or a first degree relative with breast cancer.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of women agreeing to outreach educational program | At intervention, an average of 30 minutes
  Rate of women approached who agree to enter the outreach educational program

SECONDARY OUTCOMES:
Baseline mammogram screening rate | At intervention, an average of 30 minutes
  Baseline mammogram screening rate of target population prior to enrollment in the program.
Prevalence of social barriers to cancer screening | At intervention, an average of 30 minutes
  Identify the prevalence of unique social barriers (top 3 collected will be reported) to cancer screening and prevention amongst the homeless population

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hurwitz, PhD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
This is a study to increase screening and will be studied as a population